CLINICAL TRIAL: NCT07371273
Title: Comparative Study on the Short- and Long-term Efficacy of Q-ISR, Traditional Sub-ISR, and t-ISR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Li Dawei, PhD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q-ISR
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Q-ISR (Experimental): Based on preoperative precise assessment and rectal endoscopic localization, selective resection of the internal sphincter is performed "by quadrant and quantificationally" according to the extent of lesion involvement, while striving to preserve the uninvolved quadrants and the external sphincter-levator ani complex. This aims to ensure R0 resection margins and oncological safety, while reducing the risk of low anterior resection syndrome (LARS) and accelerating the recovery of bowel control function.
  Interventions: Procedure: Quadrant-based Intersphincteric Resection

INTERVENTIONS:
Procedure: Quadrant-based Intersphincteric Resection — Q-ISR (Quadrant-based ISR): Based on preoperative precise assessment and rectal endoscopic localization, selective resection of the internal sphincter is performed "by quadrant and quantificationally" according to the extent of lesion involvement, while striving to preserve the uninvolved quadrants and the external sphincter-levator ani complex. This aims to ensure R0 resection margins and oncological safety, while reducing the risk of low anterior resection syndrome (LARS) and accelerating the recovery of bowel control function.

SUMMARY:
This comparative study evaluates the short- and long-term outcomes of Quadrant-based Intersphincteric Resection (Q-ISR) versus traditional subtotal ISR (Sub-ISR) and conventional/total ISR (t-ISR) in patients with ultra-low rectal cancer undergoing sphincter-preserving surgery, with short-term endpoints focusing on perioperative safety (operative time, blood loss, length of stay, and postoperative complications such as Clavien-Dindo grade ≥II, anastomotic leakage/stricture, and stoma reversal) and long-term endpoints assessing anorectal function recovery (LARS and Wexner scores after stoma closure) and oncologic efficacy (R0 resection, recurrence patterns, and survival outcomes), aiming to determine whether a quadrant-tailored resection strategy can better balance tumor control with anal function preservation.

ELIGIBILITY:
Inclusion Criteria:

* (1) Rectal cancer diagnosed by digital rectal examination, colonoscopy, and combined biopsy pathology. (2) The distance from the lower edge of the tumor to the dentate line is 1.5-2.0 cm. (3) Good anal function before surgery. (4) The tumor does not infiltrate the intersphincteric space. (5) The tumor length is less than 3 cm, and the proportion of the tumor occupying the intestinal lumen is less than 1/3 of the circumference. (6) American Society of Anesthesiologists (ASA) score is ≤3.

Exclusion Criteria:

* (1) Presence of distant metastasis. (2) Undifferentiated carcinoma or mucinous adenocarcinoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2029-01-07 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Wexner score | 3years
LARS scores | 3years
disease-free survival | 5years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No